CLINICAL TRIAL: NCT03273023
Title: Post-Approval Study of the PROMUS PREMIERTM Everolimus-Eluting Platinum Chromium Coronary Stent System in China
Brief Title: PROMUS PREMIER™ China Post-Approval Study
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2384
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: Promus PREMIERTM Everolimus-Eluting Platinum Chromium Coronary Stent System — Promus PREMIERTM Stent System

SUMMARY:
To compile real-world clinical outcome data for the Promus PREMIERTM Everolimus-Eluting Platinum Chromium Coronary Stent System (Promus PREMIERTM Stent System) in routine clinical practice in China.

DETAILED DESCRIPTION:
Each site will be allowed to enroll up to a maximum of 300 subjects. The scheduled follow up will occur at 30 days, 6 months, 12 months and then annually through 5 years post stent implant, for all enrolled subjects. Follow-up will be conducted via telephone contact or clinic visit

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject understands and provides written informed consent
* Subject who is clinically indicated and will have an attempt of at least one Promus PREMIERTM Stent OR Subject who is clinically indicated and was implanted with at least one Promus PREMIERTM Stent
* Subject is willing to comply with all protocol-required follow-up evaluation

Exclusion Criteria:

* Exclusion criteria are not required in the PE PREMIERTM China Post-Approval Study which is an "all comers" study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are candidates for coronary artery stenting, signed the informed consent form and eligible to receive a Promus PREMIERTM Stent System will be evaluated for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2059 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
12-month Primary Endpoint: Major Adverse Cardiac Event (MACE) rate, defined as cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR) | 12-month follow up
  The primary endpoint is the 12-month major adverse cardiac event (MACE) rate, defined as cardiac death, myocardial infarction (MI) and target vessel revascularization (TVR)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, Dr., Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided